CLINICAL TRIAL: NCT06895161
Title: Effectiveness of Home-Based Tele-Exercise vs Center-Based Exercise Programs in Patients With Prediabetes: A Comparative Study
Brief Title: Home-Based Tele-Exercise vs. Hospital-Based Exercise Programs in Patients With Prediabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Levent Karataş, PM&R Specialist M.D, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Prediabetes and exercise
Record Dates: First submitted 2025-03-24; First posted 2025-03-26 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Prediabetes; Prediabetes (Insulin Resistance, Impaired Glucose Tolerance); Telemedecine
Keywords: Prediabetes; Telemedicine; Telerehabilitation; Aerobic exercise
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: The inclusion of patients with prediabetes who have undergone an oral glucose tolerance test and have impaired fasting glucose or impaired glucose tolerance.Patients will be randomized in to 3 groups; tele-exercise,hospital based exercise or control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hospital-based exercise group (Active Comparator): Participants in the hospital-based exercise group will perform aerobic exercises under the supervision of a nurse/research doctor five days a week for three weeks in the cardiopulmonary rehabilitation unit.Aerobic exercise will include 30-minute treadmill walking at %55-75 of the maximal heart rate.At the end of three weeks the program will be terminated and a follow-up evaluation will be conducted.
  Interventions: Other: Hospital-based exercise program
- Tele-exercise group (Experimental): Participants in the tele-exercise group will be instructed to walk continuously at moderate intensity (between 55-75% of the maximum heart rate) at home or outdoors five days a week, 30 minutes each, for three weeks usuing the heart rate monitor( Polar H9).The heart rates will be monitored by providing remote access to the data of the polar. Participants will be trained in the CPET performed before treatment to walk in a way that will keep their heart rates within the desired range.During the program the researcher will call them twice a week.Phone calls will include symptom inquiry and encouraging feedback regarding exercise parameters recorded on the Polar H9. At the end of three weeks the program will be terminated and a follow-up evaluation will be conducted.
  Interventions: Other: Remotely supervised exercise at home or outdoors; Other: Phone calls with reinforcement feedback
- Control group (No Intervention): Patients will be advised to exercise at a moderate intensity (between 55-75% of maximum heart rate) five days a week, 30 minutes each, for 3 weeks, at home or outdoors as recommended for prediabetes in the routine.Participants in this group will not be monitored with Polar or any device.They will be asked to take note of the exercise they have done. Participants will be trained in the CPET performed before treatment to walk in a way to maintain their heart rate in the desired range. At the end of three weeks the program will be terminated and a follow-up evaluation will be conducted.

INTERVENTIONS:
Other: Remotely supervised exercise at home or outdoors — Aerobic exercise at home/outdoors 30 minutes each session,five days a week for three weeks using a Polar H9 heart rate monitor.
  Arms: Tele-exercise group
Other: Hospital-based exercise program — The aerobic exercise ,30 minutes each session,five days a week for three weeks at cardiopulmonary rehabilitation unit under supervision.
  Arms: Hospital-based exercise group
Other: Phone calls with reinforcement feedback — Calls twice a week that include symptom inquiries and encouraging feedback on exercise
  Arms: Tele-exercise group

SUMMARY:
This study aims to compare the effects of tele-exercise(TELE) and hospital-based exercise(HBE) on functional capacity (maximum oxygen consumption), glycemic control, quality of life and sleep quality in individuals with prediabetes. Aerobic exercise will be performed 5 days a week for 30 minutes with moderate intensity continuous walking for a total of 3 weeks.While the HBE group will the exercise program under supervision in hospital,the TELE group wil perform the exercise program at home/outdoors using Polar H9 heart rate monitor. The control group (CON) will perform the exercise program at home/outdoors without any monitoring or follow up.

DETAILED DESCRIPTION:
This prospective,randomized,controlled study aims to investigate the comparative effects of tele-exercise and hospital-based exercises on functional capacity,glycemic control,quality of life and sleep quality in individuals with prediabetes. The study is planning to be conducted between April 1, 2025 and December 15, 2025.Among those undergoing oral glucose tolerance testing, patients who meet the appropriate inclusion criteria will be included in the study.Participants will be randomized into 3 groups.Aerobic exercise in all groups will be performed 5 days a week, 30 minutes each day, for a total of 3 weeks.All groups will be initially referred to a dietitian for prediabetes.

In the HBE group patients will undergo supervised exercise sessions in the cardiac rehabilitation (CR) unit, with treadmill. Aerobic exercise will be based on the patient's peak VO2 from a baseline cardiopulmonary exercise test (CPET),aimin to achieve %55-75 of the maximum heart rate.

The TELE group will receive a home based exercise program.Aerobic exercise,such as walking,will be performed for 30 minutes,5 times a week,monitored via Polar H9 heart rate device. Patients will be asked to walk at a heart rate corresponding to 55-75% of the peak VO2 determined by CPET at baseline.Weekly remote follow ups will conduct via phonel calls to asses adherence,review heart rate data and provide encouragament.

The CON group will receive a home based exercise program too.Patients will be asked to walk at a heart rate corresponding to 55-75% of the peak VO2 determined by CPET at baseline.They will be asked to take notes after exercises. But there won't be any monitoring or follow up's to this group.

Initial and final evaluations will include CPET,2-hour glucose,Glucose area under the curve,fasting glucose,fasting insuline,Hba1c,36 Item Short-form (SF-36) Survey,Pittsburgh Sleep Quality Index,body mass index.Also at the end physical activity enjoyment scale will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the study
* ≥18 and <80 years of age
* With oral glucose tolerance test (after 75 g oral glucose) 2nd hour glucose value: 140-199 mg/dl or fasting blood glucose : 100-125 mg/dl and diagnosed as prediabetes by an endocrinologist

Exclusion Criteria:

* High physical activity: Performing ≥150 minutes of moderate-intensity exercise per week
* Using insulin or oral antidiabetics
* Presence of cardiac and physical conditions that would prevent aerobic exercise
* Presence of neurological disease with significant sensorimotor deficit
* Presence of active malignancy
* Neuropsychiatric disease or condition that may prevent cooperation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
2-hour postprandial glucose | From enrollment day to the end of the exercise program at 3 weeks.
  Plasma glucose level is measured 2 hours after the person drinks 75 g of glucose solution.(oral glucose tolerence test). Below 140 mg/dL normal, 140-199 mg/dL prediabetes, 200 mg/dL or higher indicates diabetes.
Maximum oxygen consumption (VO2max) | From enrollment day to the end of the exercise program at 3 weeks
  It is the highest amount of oxygen that patients can consume during incremental aerobic exercise and is considered the best indicator of exercise capacity.
Glucose area under the curve (AUC) | From enrollment day to the end of the exercise program at 3 weeks
  It is the value obtained by calculating the area under the curve after 75 g of Oral Glucose Tolerance Test. PG=Plasma glucose Formule is; ( PG(0) +PG(30)×2+PG(60)×3+PG(120)×2 )/4 Glucose excursion, rather than PG levels at a point, is considered to provide more information about glucose tolerance. The glucose area under the curve (AUC), which is an index of whole glucose excursion after glucose loading, has been widely used for calculating the glycemic index and for evaluating the efficacy of treatment for postprandial hyperglycemia

SECONDARY OUTCOMES:
Fasting glucose | From enrollment day to the end of the exercise program at 3 weeks.
  Fasting glucose (Fasting Blood Sugar, FBS) refers to the blood sugar level measured after at least 8-12 hours of fasting, usually in the morning before eating or drinking anything (except water). It is one of the primary tests used to screen for diabetes, prediabetes, and overall glucose metabolism.If 70-99 mg/dl normal, 100-126 mg/dl prediabetes, 126 mg/dl or higher indicates diabetes.
Fasting insuline | From enrollment day to the end of the exercise program at 3 weeks.
  It is tested in blood taken after 8-12 hours of fasting.Evaluates insulin sensitivity and resistance. High fasting insulin levels can indicate insulin resistance, where the body doesn't respond well to insulin.
36-Item Short Form Survey | From enrollment day to the end of the exercise program at 3 weeks
  It is a 36-item, patient-reported survey of patient health.It consists of eight scaled scores(vitality,physical functioning,bodily pain,general health perceptions,physical role functioning,emotional role functioning,social role functioning,mental health or emotional wellbeing) which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Pittsburgh sleep quality index | From enrollment day to the end of the exercise program at 3 weeks
  The questionnaire consists of a combination of Likerttype and open-ended questions . Respondents are asked to indicate how frequently they have experienced certain sleep difficulties over the past month and to rate their overall sleep quality.. Each component score of the questionnaire ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
Hemoglobin A1c (HbA1c) | From enrollment day to the end of the exercise program at 3 weeks
  HbA1c is a blood test that measures average blood sugar (glucose) levels over the past 2 to 3 months. It's a key marker used to diagnose and monitor diabetes and is considered one of the most reliable indicators of long-term blood glucose control.If below %5,7 normal, %5,7-6,4 prediabetes, %6,5 or higher indicates diabetes.
First Minute Heart Rate Recovery | From enrollment day to the end of the exercise program at 3 weeks
  Heart rate recovery (HRR) refers to the rate at which the heart rate declines following the cessation of exercise,reflecting the balance of autonomic nervous system function,specifically the reactivation of parasympathetic(vagal) tone and withdrawal of sympathetic stimulation.In this study HRR will be assessed as the reduction in heart rate within the first minute of recovery after maximal exertion during exercise testing.A faster HRR is generally considered a mareker of superior cardiovascular fitness and autonomic funciton.Prediabetes is associated with autonomic dysfunction.
VO2 anaerobic threshold (VO2AT) | From enrollment day to the end of the exercise program at 3 weeks
  VO2 anaerobic threshold (VO2AT) refers to the specific volume of oxygen consumed per minute (VO2) when the body reaches the anaerobic threshold (AT) during exercise. The anaerobic threshold (also known as the lactate threshold) is the point where there is a significant shift in the body's energy system from primarily aerobic metabolism (using oxygen) to anaerobic metabolism (without enough oxygen).
Physical Activity Enjoyment Scale | At the end of the exercise program at 3 weeks
  It is an 8-item scale consisting of a single dimension that evaluates positive emotions such as expected or perceived pleasure and enjoyment from physical activities. Participants are asked to indicate the extent to which they agree with each item on a seven-point scale ranging from 1 - strongly disagree to 7 - strongly agree.Higher scores indicate greater enjoyment of physical activity
Body Mass Index | From enrollment day to the end of the exercise program at 3 weeks
  Body Mass Index (BMI) is a numerical measurement that helps assess whether a person has a healthy body weight relative to their height. BMI = weight (kg) / height (m²)

CONTACTS AND LOCATIONS:
Overall Officials: Çise C Güngör, MD, Principal Investigator — Gazi University Faculty of Medicine; Nesrin Ü Demirsoy, MD, Principal Investigator — Gazi University Faculty of Medicine; Levent Karataş, MD, Principal Investigator — Gazi University Faculty of Medicine; Muhittin M Yalçın, MD, Principal Investigator — Gazi University Faculty of Medicine; Levent A Güngör, MD, Principal Investigator — Gazi University Faculty of Medicine
Locations (1):
- Gazi University Hospital,Department of Physical Medicine and Rehabilitation, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sakaguchi K, Takeda K, Maeda M, Ogawa W, Sato T, Okada S, Ohnishi Y, Nakajima H, Kashiwagi A. Glucose area under the curve during oral glucose tolerance test as an index of glucose intolerance. Diabetol Int. 2015 May 14;7(1):53-58. doi: 10.1007/s13340-015-0212-4. eCollection 2016 Mar. PMID 30603243
- [Background] Duruturk N. Telerehabilitation intervention for type 2 diabetes. World J Diabetes. 2020 Jun 15;11(6):218-226. doi: 10.4239/wjd.v11.i6.218. PMID 32547696
- [Background] Duruturk N, Ozkoslu MA. Effect of tele-rehabilitation on glucose control, exercise capacity, physical fitness, muscle strength and psychosocial status in patients with type 2 diabetes: A double blind randomized controlled trial. Prim Care Diabetes. 2019 Dec;13(6):542-548. doi: 10.1016/j.pcd.2019.03.007. Epub 2019 Apr 20. PMID 31014938
- [Background] Blioumpa C, Karanasiou E, Antoniou V, Batalik L, Kalatzis K, Lanaras L, Pepera G. Efficacy of supervised home-based, real time, videoconferencing telerehabilitation in patients with type 2 diabetes: a single-blind randomized controlled trial. Eur J Phys Rehabil Med. 2023 Oct;59(5):628-639. doi: 10.23736/S1973-9087.23.07855-3. Epub 2023 Jun 23. PMID 37350165